CLINICAL TRIAL: NCT05276323
Title: Medihoney® Derma Cream Treatment for Mild to Moderate Atopic Dermatitis in Children: an Open-label Randomized Pilot Study
Brief Title: Medihoney® Derma Cream Treatment for Mild to Moderate Atopic Dermatitis in Children Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, AMIR HOREV, Head of pediatric dermatology, Soroka University Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SorokaUMC
Record Dates: First submitted 2022-02-20; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Atopic Dermatitis
Keywords: eczema; atopic dermatitis; Medihoney dermacream
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Hydrocortisone

STUDY DESIGN:
Intervention Model Description: We conducted a randomized trial comprising children aged 2-18 diagnosed with mild to moderate AD, with an IGA of 2-3 and BSA of 1%-10%, including 30 patients, 20 using Med-D-Cream and 10 as controls using Hydrocortisone 1% cream. Patients applied creams for 2 weeks and were then followed for two weeks to measure clinical responses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medihoney Derma Cream (Experimental): Intervention group: Medihoney Derma Cream will be applied topically, twice a day, on all affected areas in the body for two weeks. Then, follow-up for two more weeks, overall participating for 4 weeks in the trial.
  Interventions: Drug: Medihoney Derma Cream
- Hydrocortisone 1% cream (Active Comparator): control group: Hydrocortisone 1% cream will be applied topically, twice a day, on all affected areas in the body for two weeks. Then, follow-up for two more weeks, overall participating for 4 weeks in the trial.
  Interventions: Drug: Hydrocortisone 1% cream

INTERVENTIONS:
Drug: Medihoney Derma Cream — applied topically, twice a day, on all affected areas in the body for two weeks.
  Arms: Medihoney Derma Cream
Drug: Hydrocortisone 1% cream — applied topically, twice a day, on all affected areas in the body for two weeks.
  Arms: Hydrocortisone 1% cream

SUMMARY:
A randomized, open-label trial comparing Medihoney Derma Cream to Hydrocortisone 1% cream. Children between the ages of 2-18 years old diagnosed with mild to moderate atopic dermatitis with an IGA (Investigator Global Assessment) score of 2-3, and a BSA (Body Surface Area) score of 1%-10% were included.

DETAILED DESCRIPTION:
A randomized trial comprising children aged 2-18 diagnosed with mild to moderate AD, with an IGA of 2-3 and BSA of 1%-10%, including 30 patients, 20 using Med-D-Cream and 10 as controls using Hydrocortisone 1% cream. Patients applied creams for 2 weeks and were then followed for two weeks to measure clinical responses and pruritus change.

ELIGIBILITY:
Inclusion Criteria:

* 2-18 years old
* mild to moderate atopic dermatitis
* an IGA score of 2-3
* BSA score of 1%-10%.

Exclusion Criteria:

* participation in any clinical trial less than 28 days before the enrollment
* AD-related systemic therapy or phototherapy within 28 days prior to the enrollment
* topical corticosteroids, calcineurin inhibitors, or PDE4 inhibitors use within 7 days prior to the enrollment

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
response rate | 1 month
  This study's primary outcome was defined as an IGA (Investigator Global Assessment) severity score of 0 or 1 with at least 1-grade reduction at visit 3. score range 0-4 (4 worse symptomes)

SECONDARY OUTCOMES:
VAS (Visual Analogue Scale) pruritis score | 1 month
  score range is 1 to 10. 1:no itch, 10:very itchy
SCORAD - (SCORing Atopic Dermatitis) | 2 weeks
  SCORAD is a clinical tool used to assess the extent and severity of eczema. range 0-103. 103- worse eczema
The Eczema Area and Severity Index (EASI) | 2 weeks
  is a validated scoring system that grades the physical signs of atopic dermatitis/eczema. The minimum EASI score is 0 and the maximum EASI score is 72 (72 worse eczema)

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No